CLINICAL TRIAL: NCT03735446
Title: Prexasertib in Combination With Mitoxantrone, Etoposide and Cytarabine (MEC) in Relapsed/Refractory Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS) - a Phase I Trial
Brief Title: Prexasertib in Combination With MEC in Relapsed/Refractory AML and High Risk MDS - a Phase I Trial
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Eric Stephen Winer, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-468
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndromes; AML; MDS; CHK1; MEC; Prexasertib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — prexasertib; Mitoxantrone; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prexasertib+MEC (Experimental): * Cytarabine is administered intravenously on days 1-5.
  * Etoposide is administered intravenously on days 1-5.
  * Mitoxantrone is administered intravenously on days 1-5.
  * Prexasertib is administered intravenously on days 1, 3, and 5.
  Interventions: Drug: Prexasertib; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: Prexasertib — Checkpoint kinase 1 (CHK1) inhibitor
  Other Names: LY2606368
Drug: Mitoxantrone — Standard chemotherapy (topoisomerase inhibitor)
  Other Names: Novantrone
Drug: Etoposide — Standard chemotherapy (topoisomerase II inhibitor)
Drug: Cytarabine — Standard chemotherapy (anti-metabolite)

SUMMARY:
This research study is studying a targeted therapy combined with chemotherapy as a possible treatment for acute myeloid leukemia (AML) or high risk myelodysplastic syndrome (MDS).

The drugs involved in this study are:

* Prexasertib (LY2606368)
* Mitoxantrone
* Etoposide
* Cytarabine

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug or combination of drugs and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved prexasertib as a treatment for any disease. Prexasertib is a checkpoint kinase 1 (CHK1) inhibitor that is being developed as a treatment for patients with advanced cancer. CHK1 inhibitors work by preventing cancer cells from being able to repair damaged DNA (one of the building blocks of a cell) which then leads to cell death.

The drugs mitoxantrone, etoposide, and cytarabine (MEC) have all been approved by the FDA. MEC is a standard chemotherapy treatment option, commonly used for AML that has not responded to other standard treatment or returned following standard treatment.

In this research study, the investigators are combining prexasertib with MEC therapy to test if it is a safe treatment for AML or MDS that has returned or not responded to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed relapsed or refractory acute myeloid leukemia (AML) or high risk myelodysplastic syndrome (MDS) diagnosed per WHO criteria.
* For refractory AML: refractory as defined per International Working Group (IWG) criteria. Refractory patients must have had ≤ 2 prior induction regimens (hydroxyurea is not considered a prior treatment regimen). "5+2" reinduction at day 14 is not considered a second regimen.
* For relapsed AML: relapse as defined by IWG criteria. Relapsed patients must be first or second relapse (hydroxyurea is not considered a prior treatment regimen).
* For patients with MDS, ≥ 10% myeloblasts in the bone marrow, and no more than 2 prior treatment regimens (hydroxyurea is not considered a prior treatment regimen).
* Patients must be medically eligible to receive mitoxantrone, etoposide, and cytarabine (MEC) therapy.
* Age ≥ 18 years
* ECOG performance status ≤ 2 (Karnofsky ≥60%)
* Patients must have adequate organ function as defined below:

  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN), OR
  * Total bilirubin ≤ 2 × institutional ULN if the participant has a history of Gilbert's syndrome.
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN, OR
  * AST(SGOT)/ALT(SGPT) ≤ 5 × institutional ULN if elevation is a result of leukemia
  * Serum creatinine ≤ 1.5 × institutional ULN, OR
  * Creatinine Clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal (calculated via the Cockcroft-Gault equation).
* Left ventricular ejection fraction (LVEF) ≥ 50% on screening echocardiogram (ECHO) or multigated acquisition scan (MUGA).
* QTcF value of ≤ 450 msec on screening electrocardiogram (ECG).
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study therapy administration. A negative serum pregnancy test is required for women of child-bearing potential.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients may have had a prior autologous or allogeneic transplant if there is at least 100 days between transplant and screening, and there is no evidence of active graft-versus-host-disease (GvHD) or ongoing requirement for immunosuppressive therapy.

Exclusion Criteria:

* Patients who have had chemotherapy, other investigational therapy, radiotherapy, or immune therapy within 2 weeks prior to the first dose of study medication. Hydroxyurea is allowed with no required washout and may be administered up to day 5 of protocol therapy.
* Patients previously treated with MEC chemotherapy.
* Patients who have received a tyrosine kinase inhibitor (TKI) within 5 half-lives of day 1.
* Patients who have had major surgery within 4 weeks prior to the first dose of study medication.
* Patients with acute promyelocytic leukemia.
* Patients with a known personal or family history of long QT syndrome.
* Patients with known CNS leukemia involvement.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to prexasertib, mitoxantrone, etoposide, or cytarabine.
* Patients with a history of a secondary malignancy, with the following exceptions:

  * Malignancies that have been curatively treated and have not recurred within the past 2 years
  * Adequately treated carcinoma in situ of any type
  * Curatively treated non-melanoma skin cancers
  * Any other malignancy that has been curatively treated with a low likelihood of recurrence as judged by the treating investigator and agreed upon with the overall principal investigator prior to study entry
  * Patients with other secondary malignancies may be allowed to enroll with agreement from the overall principal investigator.
* Uncontrolled intercurrent illness including, but not limited to: uncontrolled active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because prexasertib, mitoxantrone, etoposide, and cytarabine are anti-cancer agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study agents, breastfeeding should be discontinued if the mother is treated with prexasertib, mitoxantrone, etoposide, or cytarabine.
* Patients who are known to be seropositive for human immunodeficiency virus (HIV) or hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Up to 42 days
  Toxicities occurring following administration of protocol therapy, measured using CTCAE 5.0 criteria.

SECONDARY OUTCOMES:
Phase 2 Dose | 18 months
  Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) for the study drug combination.
Overall Response | 30 months
  Rates of complete remission (CR), complete remission with incomplete count recovery (CRi), and partial remission (PR).
Overall Survival | 30 months
  Assess the overall survival rate for the combination.
Duration of Remission | 12 months
  Time of achievement of CR or CRi to relapse, death, or 1 year (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Winer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No